CLINICAL TRIAL: NCT02649504
Title: The Study of Immunotherapy With Rituximab and Pulse Dexamethasone Followed by With Mycophenolate Mofetil or Placebo in Adult Patients With Persistent and Chronic Immune Thrombocytopenia
Brief Title: Rituximab and Dexamethasone Followed by Mycophenolate Mofetil or Placebo in Patients With Immune Thrombocytopenia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1501015858
Record Dates: First submitted 2015-12-17; First posted 2016-01-07 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab; Dexamethasone; Calcium Dobesilate; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- R+3D, MMF (Active Comparator): Rituximab will be given at the standard dose of 375mg/m2 on days 1, 8, 15, 22 of the study. Dexamethasone will be given at dose 40 mg/day on days 1-4, 15-18, and 29-32 (+/- 3 days) of the study. Mycophenolate mofetil (MMF) will be given starting on day 33, 500 mg twice daily for the first week and then escalation to 1000 mg twice daily for 24 weeks.
  Interventions: Drug: Rituximab; Drug: Dexamethasone; Drug: Mycophenolate mofetil
- R+3D, Placebo (Placebo Comparator): Rituximab will be given at the standard dose of 375mg/m2 on days 1, 8, 15, 22 of the study. Dexamethasone will be given at dose 40 mg/day on days 1-4, 15-18, and 29-32 (+/- 3 days) of the study. Placebo will be given starting on day 33, 500 mg twice daily for the first week and then escalation to 1000 mg twice daily for 24 weeks.
  Interventions: Drug: Rituximab; Drug: Dexamethasone; Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — Rituximab will be given at the standard dose of 375mg/m2 on days 1, 8, 15, 22 of the study
  Other Names: anti- cluster of differentiation antigen 20 antibody
Drug: Dexamethasone — Dexamethasone will be given at dose 40 mg/day on days 1-4, 15-18, and 29-32 (+/- 3 days) of the study.
  Other Names: Decadron, Dexasone, Diodex, Hexadrol, Maxidex
Drug: Mycophenolate mofetil — Patients allocated to the active drug arm will be given Mycophenolate mofetil starting on day 33, 500 mg twice daily for the first week and then escalation to 1000 mg twice daily for 24 weeks.
  Other Names: Cellcept
  Arms: R+3D, MMF
Drug: Placebo — Patients allocated to the placebo arm will be given placebo starting on day 33, 500 mg twice daily for the first week and then escalation to 1000 mg twice daily for 24 weeks.
  Other Names: inactive drug, fake pill
  Arms: R+3D, Placebo

SUMMARY:
The investigators will attempt to further increase the cure rate of ITP with medical therapy by providing maintenance therapy with Mycophenolate mofetil (MMF) to persistent/chronic ITP patients after treating them with induction therapy combining rituximab and dexamethasone. The investigators will randomly assign patients to MMF versus placebo in order to demonstrate safety (e.g., for infectious risk) and efficacy (platelet counts stably >50x109/L more than 1 year off therapy).

DETAILED DESCRIPTION:
There are significant numbers of Immune Thrombocytopenia (ITP) patients 18 years of age or older who relapse and become refractory after short responses to initial therapy (usually corticosteroids) or who do not respond at all. Despite a variety of available therapies, there are patients with persistently low platelet counts and bleeding complications, and there are other patients who suffer from the side effects of current treatments. Thus, there still remains an unmet need for better treatments in these patients. Based on the investigators' experience, it is expected that most of ITP patients treated with intensive induction therapy (Dexamethasone combined with rituximab, R+3D) will increase their platelet counts, and the investigators hope that a further 6-month course of Mycophenolate Mofetil will help patients to maintain continuous response and even achieve a cure of ITP. The increase in platelet count will likely result in a decreased risk for bleeding and better health-related quality of life. In addition, responders potentially will be able to stop concomitant ITP medications and will not suffer from adverse events of various ITP therapies and will avoid undergoing splenectomy.

This multi-center, randomized study will help physicians determine the best treatment option for ITP patients and may help to establish a new standard of care.

The knowledge to be gained is that of:

1. whether R+3D and placebo confirms the previous data on R+3D
2. whether R+3D + MMF increases the cure rate of ITP
3. whether R+3D + MMF increases the risk of serious infections

The investigators do not believe that the triple therapy will result in a high rate of serious infections based on the past track record of R+3D and of MMF in combination with other stronger immunosuppressive medications such as cyclosporine and tacrolimus. Therefore the risk will be limited and worth the increase in cure rate that we expect.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, greater than 18 years old
* Signed written informed consent obtained prior to study entry
* Immune Thrombocytopenia according to the American Society of Hematology guidelines, with other potential causes of thrombocytopenia excluded, platelets less than 30 x 109/L at study entry
* Have adequate renal and hepatic function (creatinine and bilirubin less than 2 x Upper Limit of Normal (ULN), aspartate aminotransferase and alanine aminotransferase less than 3 x ULN)
* No significant cytopenias (hemoglobin greater than10 g/dL without ongoing transfusional support, absolute neutrophil count greater than 1.0 x109/L at study entry).
* If on corticosteroids, receiving less than or equal to 20 mg/day prednisone (or equivalent) with no change of dose for at least 2 weeks prior to study entry. No more than two 4-day courses of Dexamethasone prior to study entry. If on danazol, no change of dose for at least 2 weeks prior to study entry. (Thrombopoietin receptor agonist treatment will be allowed until the end of 8th week on study if started prior to study entry)
* No treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half-lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study
* No prior treatment with anti-B-lymphocyte antigen cluster of differentiation antigen 20 monoclonal antibody at a total dose greater than 375mg/m2
* Screen for Hepatitis B and be negative for Hepatitis B surface antigen
* Human Immunodeficiency Virus negative
* No history of active hepatitis C infection or a past history hepatitis C (confirmed by negative anti- Hepatitis C Virus Antibody)
* No past history of tuberculosis
* No chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, or chronic chest infection with bronchiectasis
* No current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease meeting laboratory threshold limits per investigator discretion)
* No significant concurrent, uncontrolled medical condition including but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease, which in the opinion of the investigator may represent a risk for the patient. Have no past or current malignancy for 3 years (excluding nonmelanoma skin cancers, e.g., basal cell carcinoma (BCC) and carcinoma in situ of the cervix)
* Women of childbearing potential must have a negative pregnancy test at screening
* No history of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae.
* No history of venous or arterial thromboembolism in the past year.
* No clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities

Exclusion Criteria:

* Pregnant or lactating women
* Women of childbearing potential and fertile men who are not practicing or who are unwilling to practice birth control while enrolled in the study or until at least 6 months after treatment. Women of childbearing potential must have a negative pregnancy test at screening. Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy will be excluded from study. Adequate contraception is defined as intrauterine device, tubal sterilization, patient's partner had a vasectomy or total abstinence. Other contraceptive methods include hormonal contraceptive pills. Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy will be excluded from the study as well.
* Immunosuppressive agents or ITP treatments or other experimental treatments for ITP within 2 weeks. Intravenous Immunoglobulin, anti-Rh(D) prior to first day of rituximab treatment
* Splenectomy or any other surgery within 4 weeks
* Red blood cell transfusion or hospitalization for bleeding within 4 weeks
* Concomitant anticoagulation therapy (warfarin, enoxaparin, dabigatran, rivaroxaban, apixaban, fondaparinux) or any platelet aggregation inhibitors including aspirin and clopidogrel (until platelets stable greater than 100x109/L)
* New York Heart Classification III or IV heart disease. Other severe cardiovascular or cardiopulmonary disease, including chronic obstructive pulmonary disease
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-01 (Estimated); Primary Completion 2016-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a platelet count greater or equal to 50,000 for 5 of 6 platelet counts in the second half of second year (month 19 to month 24) with no rescue therapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James B. Bussel, M.D, Principal Investigator — Weill Medical College of Cornell University

REFERENCES:
- [Background] Bussel JB, Lee CS, Seery C, Imahiyerobo AA, Thompson MV, Catellier D, Turenne IG, Patel VL, Basciano PA, Elstrom RL, Ghanima W. Rituximab and three dexamethasone cycles provide responses similar to splenectomy in women and those with immune thrombocytopenia of less than two years duration. Haematologica. 2014 Jul;99(7):1264-71. doi: 10.3324/haematol.2013.103291. Epub 2014 Apr 18. PMID 24747949
- [Background] Stasi R, Pagano A, Stipa E, Amadori S. Rituximab chimeric anti-CD20 monoclonal antibody treatment for adults with chronic idiopathic thrombocytopenic purpura. Blood. 2001 Aug 15;98(4):952-7. doi: 10.1182/blood.v98.4.952. PMID 11493438
- [Background] Stasi R, Stipa E, Forte V, Meo P, Amadori S. Variable patterns of response to rituximab treatment in adults with chronic idiopathic thrombocytopenic purpura. Blood. 2002 May 15;99(10):3872-3. doi: 10.1182/blood-2002-02-0392. No abstract available. PMID 12014370
- [Background] Patel VL, Mahevas M, Lee SY, Stasi R, Cunningham-Rundles S, Godeau B, Kanter J, Neufeld E, Taube T, Ramenghi U, Shenoy S, Ward MJ, Mihatov N, Patel VL, Bierling P, Lesser M, Cooper N, Bussel JB. Outcomes 5 years after response to rituximab therapy in children and adults with immune thrombocytopenia. Blood. 2012 Jun 21;119(25):5989-95. doi: 10.1182/blood-2011-11-393975. Epub 2012 May 7. PMID 22566601
- [Background] Zaja F, Baccarani M, Mazza P, Bocchia M, Gugliotta L, Zaccaria A, Vianelli N, Defina M, Tieghi A, Amadori S, Campagna S, Ferrara F, Angelucci E, Usala E, Cantoni S, Visani G, Fornaro A, Rizzi R, De Stefano V, Casulli F, Battista ML, Isola M, Soldano F, Gamba E, Fanin R. Dexamethasone plus rituximab yields higher sustained response rates than dexamethasone monotherapy in adults with primary immune thrombocytopenia. Blood. 2010 Apr 8;115(14):2755-62. doi: 10.1182/blood-2009-07-229815. Epub 2010 Feb 3. PMID 20130241